CLINICAL TRIAL: NCT01538862
Title: Efficacy of Granulocyte Colony Stimulating Factor (GCSF) In Patients With Dystrophic Epidermolysis Bullosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Haydar Frangoul, Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICCNCPED1210
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Granulocyte Colony Stimulating Factor (GCSF) (Experimental): GCSF 10mcg/kg/d subcutaneously (SQ) for 7 days
  Interventions: Drug: Granulocyte Colony Stimulating Factor (GCSF)

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor (GCSF) — G-CSF 10mcg/kg/d SQ for 7 days

SUMMARY:
This is a feasibility study to see if Granulocyte Colony Stimulating Factor (GCSF) is effective as a treatment of Dystrophic Epidermolysis Bullosa (EB). Patients will receive one course of treatment with the study drug. The course will be 7 days in length. After receiving GCSF, patients will be followed at 7 and 30 days following the discontinuation of the drug. Thirty day follow up can be done via telephone communication with the patient or family.

DETAILED DESCRIPTION:
Each patient will be given 10 micrograms per kilogram per day of G-CSF subcutaneously for 6 consecutive days. On day 7 each patient will be seen and evaluated in the same manner as on day 0. Patients or their parents (if children are too young to reliably respond themselves) will also be asked to rate the following via a visual analog scale of 1-9- oral pain, pruritus, oral pain, swallowing, and overall sense of well-being. A telephone follow-up will be conducted on all patients 28 days after G-CSF so as to evaluate if the effect noted on day 7 was sustained.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must have the diagnosis of severe generalized recessive dystrophic EB (formerly known as Hallopeau-Siemens RDEB) confirmed by clinical criteria and either of the following:

  1. transmission electron microscopy
  2. immunofluorescence antigenic mapping and type VII collagen monoclonal antibody staining
  3. COL7A1 mutational analysis

Exclusion Criteria:

* The patient must not have a history of squamous cell carcinoma or any internal malignancy.
* Female patients who are pregnant.
* Patients with active signs and symptoms of infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Frangoul, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Granulocyte Colony Stimulating Factor (GCSF): GCSF 10mcg/kg/d SQ for 7 days
  Granulocyte Colony Stimulating Factor (GCSF): G-CSF 10mcg/kg/d SQ for 7 days
Period: Overall Study
Arm/Group | Granulocyte Colony Stimulating Factor (GCSF)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Granulocyte Colony Stimulating Factor (GCSF)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Active Blisters and in Total Blister/Erosion Counts
Description: Percent change of active blisters and in total blister/erosion counts from baseline to 7 days
Time Frame: 7 days
Population: Time frame was originally entered as 30 days. This was not consistent with the protocol which listed a 7 day time frame for this Outcome
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Granulocyte Colony Stimulating Factor (GCSF): GCSF 10mcg/kg/d subcutaneously for 7 days
  Granulocyte Colony Stimulating Factor (GCSF): G-CSF 10mcg/kg/d subcutaneously for 7 days
Arm/Group | Granulocyte Colony Stimulating Factor (GCSF)
Number analyzed (Participants) | 7
percent change | -29.6 (30.3)
Statistical Analysis 1: Comparison: Granulocyte Colony Stimulating Factor (GCSF); Test type: Superiority; p = 0.82, Regression, Linear

2. Secondary Outcome: Surface Area of Nonhealing Erosions
Description: Change in surface area of one or two nonhealing erosions
Time Frame: 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Granulocyte Colony Stimulating Factor (GCSF)
Number analyzed (Participants) | 7
percentage change | -35.3 (100.8)

3. Secondary Outcome: Overall Improved Symptomatology
Description: Overall clinical improvement in symptomatology and/or findings, as assessed by either the patient or parent. This would include decrease in the number and size of blister and erosions, decreased pain, improved comfort of the patient.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Granulocyte Colony Stimulating Factor (GCSF)
Number analyzed (Participants) | 7
Participants | 6

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Granulocyte Colony Stimulating Factor (GCSF)
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes